CLINICAL TRIAL: NCT06030726
Title: Nationwide Utilization of Danish Government Electronic Letter System for Confirming the Effectiveness of Behavioral Nudges in Increasing InFLUenza Vaccine Uptake Among Older Adults
Acronym: NUDGE-FLU-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NUDGE-FLU-2
Record Dates: First submitted 2023-08-31; First posted 2023-09-11 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Influenza; Behavior and Behavior Mechanisms
Keywords: Influenza; Vaccination; Nudging; Behavioral Science
MeSH Terms: conditions — Influenza, Human; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Usual Care (No Intervention): No letter
- Standard Letter (Experimental): This group will receive a standard letter on the benefits of influenza vaccination without behavioral economic enhancement
  Interventions: Behavioral: Behavioral Economic Principles
- Repeated Letter (Experimental): The standard letter sent out two times instead of once
  Interventions: Behavioral: Behavioral Economic Principles
- Cardiovascular Gain-Framing Letter (Experimental): Text added to the standard letter highlighting potential cardiovascular benefits of influenza vaccination
  Interventions: Behavioral: Behavioral Economic Principles
- Respiratory Gain-Framing Letter (Experimental): Text added to the standard letter highlighting potential respiratory disease-related benefits of influenza vaccination
  Interventions: Behavioral: Behavioral Economic Principles
- Implementation Intention Prompt Letter (Experimental): Implementation intention prompt added to the standard letter
  Interventions: Behavioral: Behavioral Economic Principles
- Loss-Framing Letter (Experimental): Text added to the standard letter highlighting potential risks of not receiving influenza vaccination
  Interventions: Behavioral: Behavioral Economic Principles

INTERVENTIONS:
Behavioral: Behavioral Economic Principles — The control arm will receive no letter to reflect the background vaccination uptake. Intervention arms will test the effects of different letters developed using behavioral economic principles.
  Arms: Cardiovascular Gain-Framing Letter; Implementation Intention Prompt Letter; Loss-Framing Letter; Repeated Letter; Respiratory Gain-Framing Letter; Standard Letter

SUMMARY:
In randomized clinical trials and observational studies, influenza vaccination has been shown to be effective in reducing influenza-related illness, hospitalizations, cardiovascular events, and mortality in select populations. However, the real-world effectiveness of influenza vaccination is limited by its uptake. Conducted during the 2022/2023 influenza season, the first NUDGE-FLU trial demonstrated the effectiveness of two electronic behavioral nudging letter strategies in increasing influenza vaccination rates among older adults in Denmark - a letter highlighting potential cardiovascular benefits of vaccination and a standard informational letter sent at baseline and repeated at day 14. This present study will once again investigate whether digital behavioral nudges delivered via the official, mandatory Danish electronic letter system can increase influenza vaccine uptake among older adults including whether the effectiveness of previously successful strategies can be confirmed during a subsequent influenza season.

DETAILED DESCRIPTION:
The study is a prospective, randomized, open-label implementation trial. The study population will consist of persons aged >=65 years at January 15, 2024 - this age group is eligible for free-of-charge influenza vaccination in the official Danish vaccination program. Subjects will be identified through Danish nationwide health registries including the Danish Civil Registration System. Individuals will be randomized to 1 of 7 arms (1 usual care arm and 6 intervention arms) with each testing different nudging strategies employing various behavioural economic principles. The interventions will be delivered through the official, mandatory Danish electronic letter system. All subject data will be retrieved from the Danish nationwide registries with the exception of information on intervention allocation. Endpoints will be retrieved at prespecified dates using prespecified search algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=65 years at January 15, 2024 (eligible for free-of-charge influenza vaccination in the Danish public health system)
2. Access to the official, mandatory Danish electronic mailbox system

Exclusion Criteria:

1. Persons living in nursing homes (approximated as any person living at an address with >=6 inhabitants aged 80 years and above)
2. Known to have already scheduled influenza vaccination appointment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 881373 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who received an influenza vaccine | Up to 3 months

SECONDARY OUTCOMES:
Time from intervention delivery to influenza vaccination | Up to 3 months

OTHER OUTCOMES:
Number of participants with laboratory-confirmed influenza | Up to 8 months
Number of participants with a hospitalization for influenza or pneumonia | Up to 8 months
Number of participants with a hospitalization for any respiratory disease | Up to 8 months
Number of participants with a hospitalization for any cardio-respiratory disease | Up to 8 months
Number of participants with a hospitalization for any cardiovascular disease | Up to 8 months
Number of participants with any hospitalization | Up to 8 months
Total number of hospitalizations (first and recurrent) | Up to 8 months
All-cause mortality | Up to 8 months
Composite of incident heart failure, heart failure hospitalization, or cardiovascular death | Up to 8 months
Composite of myocardial infarction, stroke, or cardiovascular death | Up to 8 months
Composite of myocardial infarction, coronary revascularization, stroke, or cardiovascular death | Up to 8 months
Number of participants with incident heart failure or heart failure hospitalization | Up to 8 months
Total number of heart failure events (incident heart failure and first and recurrent heart failure hospitalizations) | Up to 8 months
Cardiovascular death | Up to 8 months
Number of participants with myocardial infarction | Up to 8 months
Number of participants with coronary revascularization | Up to 8 months
Number of participants with stroke | Up to 8 months
Number of participants with incident atrial fibrillation or atrial fibrillation hospitalization | Up to 8 months
Number of contacts to general practitioner (excluding vaccination visit) | Up to 8 months
Number of participants with laboratory-confirmed COVID-19 | Up to 8 months
Number of participants with a hospitalization for COVID-19 | Up to 8 months
Number of participants who received a COVID-19 vaccine | Up to 3 months
Number of participants who filled a prescription for any guideline-directed medical therapy for heart failure | Up to 8 months
Total number of filled prescriptions for guideline-directed medical therapy for heart failure | Up to 8 months
Number of participants who filled a prescription for a sodium-glucose cotransporter 2 inhibitor or glucagon-like peptide 1 receptor agonist | Up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, MSc, MPH, PhD, Principal Investigator — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.

REFERENCES:
- [Derived] Bhatt AS, Johansen ND, Vaduganathan M, Modin D, Pareek M, Chatur S, Claggett BL, Janstrup KH, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Dueger EL, Samson S, Loiacono MM, Harris RC, Kober L, Solomon SD, Martel CJ, Sivapalan P, Jensen JUS, Biering-Sorensen T. Electronic Nudges and Influenza Vaccination Among Patients With a History of Myocardial Infarction: Insights From 3 Nationwide Randomized Clinical Trials. JAMA Cardiol. 2025 Jan 1;10(1):78-86. doi: 10.1001/jamacardio.2024.4648. PMID 39550717
- [Derived] Johansen ND, Vaduganathan M, Bhatt AS, Modin D, Chatur S, Claggett BL, Janstrup KH, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Martel CJ, Krause TG, Biering-Sorensen T. Electronic nudges for sustained influenza vaccination uptake in older adults: the nationwide randomized NUDGE-FLU-2 trial. Nat Med. 2024 Nov;30(11):3142-3149. doi: 10.1038/s41591-024-03202-4. Epub 2024 Aug 30. PMID 39215149
- [Derived] Johansen ND, Vaduganathan M, Bhatt AS, Modin D, Chatur S, Claggett BL, Janstrup KH, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Martel CJ, Krause TG, Biering-Sorensen T. Rationale and design of NUDGE-FLU-CHRONIC and NUDGE-FLU-2: Two nationwide randomized trials of electronic nudges to increase influenza vaccination among patients with chronic diseases and older adults during the 2023/2024 influenza season. Am Heart J. 2024 Jun;272:23-36. doi: 10.1016/j.ahj.2024.03.003. Epub 2024 Mar 7. PMID 38460754